CLINICAL TRIAL: NCT03383354
Title: Examining the Link Between Clinical and Physiological Sleep Data and Health-related Outcomes
Brief Title: The Link Between Clinical and Physiological Sleep Data and Health-related Outcomes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Institute for Clinical Evaluative Sciences (Other); Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 095-2016
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Sleep Apnea Syndromes; Cardiovascular Diseases; Sleep Initiation and Maintenance Disorders; Nocturnal Myoclonus Syndrome; Hospitalizations; Mortality; Cancer
MeSH Terms: conditions — Sleep Apnea Syndromes; Cardiovascular Diseases; Sleep Initiation and Maintenance Disorders; Nocturnal Myoclonus Syndrome; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sleep-related disturbances (exposure) — Sleep-related disturbances such as sleep-disordered breathing (e.g. sleep apnea), sleep fragmentation, abnormal sleep architecture, and periodic limb movements (PLMs)

SUMMARY:
Emerging evidence suggests that sleep-related disturbances such as sleep-disordered breathing (e.g. sleep apnea), sleep fragmentation, abnormal sleep architecture, and periodic limb movements (PLMs) are closely linked with adverse health outcomes such as cardiovascular events, hospital admissions and mortality. However, data supporting some of these associations is inconclusive. The Sunnybrook Health Sciences Centre sleep clinic has collected a detailed set of physiological variables from adults who underwent daytime and overnight sleep studies at the Sunnybrook Health Sciences Centre Sleep Laboratory from 2004 till present. Data exists on more than 5,000 subjects with various disturbances of sleep. The investigators plan to link the Sunnybrook Sleep Laboratory data with various health administrative databases based at the Institute for Clinical Evaluative Sciences (ICES). The primary objective of this study is to determine whether the presence of various findings on polysomnography (e.g. obstructive sleep apnea, sleep structure / fragmentation, physiological characteristics such as arousals and periodic limb movements in sleep) are associated with different adverse health outcomes such as cardiovascular events, cancer, depression, hospital admissions, emergency department visits and mortality.

DETAILED DESCRIPTION:
The investigators will conduct a population-based cohort study using linked provincial health administrative data (based at ICES) and clinical sleep data from the Sunnybrook Health Sciences Centre Sleep Laboratory.

ICES holds an individual-level, longitudinal, coded, linkable and secure and privacy protected health databases on most publicly funded health services for the Ontario population eligible for universal health coverage since 1991 (http://www.ices.on.ca/Data-and-Privacy/ICES-data). The records in ICES data include information on physician claims submitted to the Ontario Health Insurance Plan, discharge summaries of emergency department visits and hospital stays and for those 65 years and older medical drug claims to the Ontario Drug Benefit Program. These databases will be linked using unique encoded identifiers and analysed at ICES.

In Ontario, details on physician and hospital services are captured in several health administrative databases; of these databases, the investigators plan to use the following datasets among others: (i) the Ontario Health Insurance Plan (OHIP) physician services database; (ii) the Canadian Institute for Health Information Discharge Abstract Database; (iii) the Ontario Registered Persons Database; (iv) Ontario Registrar General - Death (Vital Stats); and (v) the Ontario Stroke Registry.

ICES is a prescribed entity under section 45 of Ontario's Personal Health Information Protection Act (PHIPA). Section 45 is the provision that enables analysis and compilation of statistical information related to the management, evaluation and monitoring of, allocation of resources to, and planning for the health system. Section 45 authorizes health information custodians to disclose personal health information to a prescribed entity, like ICES, without consent for such purposes.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients who underwent a daytime or night-time sleep study at the Sunnybrook Health Sciences Centre Sleep Laboratory

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will retrospectively analyze data from patients who underwent a daytime or night-time sleep study at the Sunnybrook Health Sciences Centre Sleep Laboratory. We plan to link sleep-related data using patients' last and first name, date of birth, gender and postal code, to health administrative data housed at the Institute for Clinical Evaluative Sciences (ICES). The full date of birth and full postal code are required to establish precise linkages with ICES outcomes data.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Composite: cardiovascular events and mortality | From initial diagnostic sleep study to March 2018
  Defined from health administrative data using validated case definition

SECONDARY OUTCOMES:
Separate components of the composite outcome | From initial diagnostic sleep study to March 2018
  Defined from health administrative data using validated case definition
Incident and prevalent cancer | From initial diagnostic sleep study to March 2018
  Defined from health administrative data using validated case definition
Hospitalizations | From initial diagnostic sleep study to March 2018
  Defined from health administrative data using validated case definition
Emergency department visits | From initial diagnostic sleep study to March 2018
  Defined from health administrative data using validated case definition

CONTACTS AND LOCATIONS:
Overall Officials: Tetyana Kendzerska, MD PhD, Principal Investigator — University of Ottawa
Locations (1):
- Dr. Mark I. Boulos - Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Kendzerska T, Murray BJ, Gershon AS, Povitz M, McIsaac DI, Bryson GL, Talarico R, Hilton J, Malhotra A, Leung RS, Boulos MI. Polysomnographic Assessment of Sleep Disturbances in Cancer Development: A Historical Multicenter Clinical Cohort Study. Chest. 2023 Aug;164(2):517-530. doi: 10.1016/j.chest.2023.03.006. Epub 2023 Mar 11. PMID 36907376